CLINICAL TRIAL: NCT02045329
Title: Impact of Mupirocin Decolonization on the Nasal Microbiome
Status: Terminated | Type: Observational
Why Stopped: Logistically unable to recruit subjects
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: COMIRB 13-1513; Grant funding (Other Grant/Funding Number: VA Merit Review Grant I01BX007080)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-05

CONDITIONS: Nasal Colonization With Staph Aureus
Keywords: Staphylococcus aureus, mupirocin, decolonization
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Staphylococcus aureus nasal carriers: Patients who are treated with mupirocin to clear nasal colonization with Staphylococcus aureus

SUMMARY:
The normal bacteria that inhabit the human nose, also known as the nasal microbiome, may serve as a host defense mechanism against colonization and infection by Staphylococcus aureus, including methicillin resistant S. aureus (MRSA). Mupirocin is a topical antibacterial agent that may be used to clear nasal colonization with S. aureus, and reduce risk of S. aureus infection. The impact of mupirocin on the normal nasal microbiome is not known. We hypothesize that the nasal microbiome is changed by mupirocin. Our study aims to define the nasal microbiome before and after decolonization therapy with mupirocin.

DETAILED DESCRIPTION:
A. Outcome Measures: This is essentially a descriptive study. We will define the nasal microbiota before and after decolonization therapy with mupirocin.

B. Description of Population to be Enrolled: Patients at VA-Denver who are starting a course of nasal mupirocin therapy for S. aureus decolonization will be enrolled. The common indications for decolonization therapy are preparation for joint replacement surgery and to facilitate removing patient from isolation for a prolonged stay on the rehabilitation service. Written informed consent will be obtained.

C. Study design and research methods: A nasal swab will be obtained just prior to initiation of mupirocin therapy, within 48 hours of the completion of mupirocin therapy, one week, two weeks, four weeks, eight weeks, and 16 weeks following the completion of mupirocin therapy. The swab will be inserted into one nare and rotated for 3 seconds. The procedure will be repeated on the other nare. The two heads will be refrigerated immediately, and held at 2-5o C until they can be placed into sterile micro tubes for storage at -80o C. A separate swab will be passed through the mouth and rubbed over the tonsils and posterior oropharynx , and stored in the same fashion.

Broad-Range PCR and High throughput DNA Sequencing PCR amplification and sequencing of rRNA genes will follow our previously published protocol (13). In brief, DNA lysates are subjected to PCR with pan-bacterial 16S rDNA rDNA primers, which yields libraries of PCR amplicons representative of all bacteria or fungi in a specimen (14). Triplicate PCR reactions will be performed and amplicons pooled for each sample. Poisoning controls spiked with bacterial (e.g. Bacillus subtilis) genomic DNA will be assayed to detect the presence of PCR inhibitors in template DNA preparations; although not typically a problem with nasal swabs, inhibitory samples will be purified by ethanol precipitation and then resubmitted for PCR. PCR amplicon libraries will be sequenced using the high-throughput Illumina MiSeq personal sequencing platform. which is available through the University of Colorado's Division of Infectious Diseases. This platform can generate 5-20x106 DNA sequences in a single instrument run with mean read lengths ~450 nts. The primers used for broad-range PCR include unique barcoded sequences in order to simultaneously sequence multiple amplicon libraries in a single instrument run (15). We will construct and sequence libraries from 100 specimens (50 persistent MRSA carriers [cases] and 50 non-carriers [controls]) to a depth of >50,000 high-quality sequencing reads per specimen. Our preliminary study indicates that this depth of coverage will represent a complete survey of the nares microbiota for each specimen.

Sequence Analysis Microbes present in specimens will be identified through use of the Naïve Bayesian Classifier Tool (16) of the Ribosomal Database Project (17). To reduce the overall complexity of the datasets, similar rDNA sequences will be clustered into operational taxonomic units (OTUs) by clustering sequences based on taxonomic assignments. Data matrices are then assembled that tabulate the frequency of each OTU in a sample. Sampling coverage for each amplicon library will be estimated (18-20) and additional sequences screened if coverage is less than 95%. All sequences will be deposited into GenBank for public use.

Validation of candidate microorganisms Microbes identified through broad-range rDNA analysis as potentially impacting S. aureus colonization will be further evaluated based on targeted QPCR measurements. Based on our preliminary results and previously published studies that suggest their interference with S. aureus growth, both S. epidermidis, (femA) and Corynebacterium spp., (rpoB PCR) will be enumerated by Q-PCR (Table, below). Primer sets for Q-PCR assays of novel microbial groups will be designed for detection of rDNA operons (i.e. 16S-ITS-23S genes) through the ARB software package (21). In the case of previously recognized microbial groups and/or species, PCR primer sets may be identified by literature search.

ELIGIBILITY:
Inclusion Criteria: - Patients at VA-ECHCS who are starting a course of nasal mupirocin therapy for S. aureus decolonization

Exclusion Criteria:

Age < 18 years Pregnant women Prisoners Decisionally challenged subjects

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated with mupirocin to clear nasal colonization with Staphylococcus aureus
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

PRIMARY OUTCOMES:
Nasal microbiome changes with mupirocin | 16 weeks
  This is a descriptive study. We will define the nasal microbiota before and after decolonization therapy with mupirocin.

SECONDARY OUTCOMES:
Recurrence of S. aureus colonization | 16 weeks
  We will look at differences in the nasal microbiome of subjects who realpse with colonization and those who remain free of S. aureus colonization.

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Bessesen, MD, Principal Investigator — Veterans Affairs Eastern Colorado Healthcare System
Locations (1):
- Veterans Affairs Eastern Colorado Healthcare System, Denver, Colorado, United States

REFERENCES:
- [Background] Frank DN, Feazel LM, Bessesen MT, Price CS, Janoff EN, Pace NR. The human nasal microbiota and Staphylococcus aureus carriage. PLoS One. 2010 May 17;5(5):e10598. doi: 10.1371/journal.pone.0010598. PMID 20498722